CLINICAL TRIAL: NCT04963569
Title: Mechanistic Inflammatory Sub-study Embedded Within the Albumin vs Balanced Crystalloid Trial
Acronym: MIS-ABC Sepsis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Royal College of Emergency Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: AC21050; G/2021/1 (Other Grant/Funding Number: Royal College of Emergency Medicine); 301333 (Other: IRAS (England)); 300332 (Other: IRAS (Scotland))
Record Dates: First submitted 2021-06-10; First posted 2021-07-15 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Sepsis
Keywords: sepsis; infection; inflammation; cytokine; interleukin; intravenous; fluids; resuscitation; albumin; crystalloid
MeSH Terms: conditions — Sepsis; Infections; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4ml EDTA Tube - Whole blood through venepuncture 2.5ml PAXGene Tube - Whole blood through venepuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Albumin: Participants enrolled in the ABC Sepsis trial who have been randomised to 5% Human Albumin Solution as the sole resuscitative fluid in the first 6 hours.
- Balanced Crystalloid: Participants enrolled in the ABC Sepsis trial who have been randomised to Balanced Crystalloid as the sole resuscitative fluid in the first 6 hours.

SUMMARY:
MIS-ABC Sepsis is a sub-study looking to understand how the immune response in patients with infection changes during the early stages of the illness, as well as after intravenous fluid treatment. Participants in the main trial will be given one of two types of fluid (Human Albumin Solution (HAS) and Balanced Crystalloid) via a drip when they present to the hospital with severe infection (sepsis). The main trial is assessing which fluid is better, and we are going to take three blood samples around the time people come to hospital to see what happens to their immune system as a result of the infection and fluid treatment. We hope our findings will explain why one fluid might be better than another. It may also give us an important information about whether we can predict which people might get sicker despite treatment.

DETAILED DESCRIPTION:
MIS-ABC Sepsis is linked to the ABC-Sepsis trial, a pilot feasibility trial recruiting patients with community acquired infection/sepsis with a NEWS2 score of five or more and randomising the participants to receiving either balanced crystalloid or 5% HAS as the intravenous resuscitation fluid up to six hours after randomisation.

MIS-ABC Sepsis will take serial blood samples from a small number of these participants, at hospital presentation and at two further points early during the patient's admission, to allow analysis of how inflammation changes during their course of illness. Investigating temporal change and differences between treatment arms of the main study will allow a nuanced analysis of the interplay between severity of illness, physiological changes over time and any potential differences between fluid treatment arm.

This is a prospective observational study enrolling patients randomised to the ABC Sepsis study. Centres for this trial will be selected from UK NHS hospitals who are recruiting to the main ABC Sepsis study. Participants will be recruited as soon as possible, and up to 12 hours after presentation to the Emergency Department, Surgical Assessment Unit or Medical Admissions Unit.

The treatment phase of the main study spans 6 hours following randomisation, with the follow up period extending to 90 days. This sub-study requires three blood samples: immediately after enrolment, at approximately 12 and 24 hours thereafter. The follow up period similarly extends to 90 days, using routine data from the medical records for follow up.

ELIGIBILITY:
Inclusion Criteria:

* Able to obtain informed consent
* Eligible for and randomised into the ABC Sepsis trial

Exclusion Criteria:

* Excluded from the ABC Sepsis trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals presenting to the Emergency Department, Acute Medical Unit or Surgical Admission Unit.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Gray, MD, Study Director — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share study day according to the FAIR principles, after agreement with the study sponsor policies.

REFERENCES:
- See also: ABC Sepsis Trial Registration — https://www.clinicaltrials.gov/ct2/show/NCT04540094
- See also: Study Webpage — https://www.emergeresearch.org/trial/mis-abc-sepsis/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Albumin | Balanced Crystalloid
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albumin | Balanced Crystalloid | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 10 | 10 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis.
Description: Exploratory analysis to map mechanistic inflammatory response over time: 0, 12 and 24 hours. As the analysis is exploratory, there is no defined limit to cell types or cytokines measured.
  Cytokines measured: tumour necrosis factor alpha (TNF-alpha), interleukin 6 (IL-6), granulocyte-macrophage colony-stimulating factor (GM-CSF), C-X-C motif chemokine ligand 10 (CXCL10), interleukin 5 (IL-5), interferon alpha 2 (IFN-a2), interleukin 4 (IL-4), C-C motif chemokine ligand 3 (CCL3), interleukin 10 (IL-10), interleukin 12p70 (IL-12p70), C-C motif chemokine ligand 20 (CCL20), interferon gamma (IFN-gamma), C-X-C motif chemokine ligand 8 (CXCL8), and C-C motif chemokine 4(CCL4).
  This outcome measure describes the number of participants who were eligible for inclusion in the exploratory analysis described above and in later outcomes.
  Units: number of participants eligible for inclusion in comparison.
Time Frame: At presentation, 12 and 24 hours.
Population: Non-numerical outcome; all participants included in analysis.
Measure: Number; unit: participants
Groups:
- Albumin: 5% HAS
- Crystalloid: Balanced crystalloid
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
participants | 14 | 12

2. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. TNF-alpha at Presentation
Description: Exploratory analysis to map mechanistic inflammatory response. Comparison of mean cytokine concentrations between allocation arms. Comparing at presentation.
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 18.3 (18.9) | 8.7 (14.9)

3. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. TNF-alpha at 12 Hours
Description: Exploratory analysis to map mechanistic inflammatory response. Comparison of mean cytokine concentrations between allocation arms. Comparing at 12 hours.
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 15.4 (14.0) | 6.6 (6.8)

4. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. TNF-alpha at 24 Hours
Description: Exploratory analysis to map mechanistic inflammatory response. Comparison of mean cytokine concentrations between allocation arms. Comparing at 24 hours.
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 16.5 (14.2) | 7.3 (10.3)

5. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. GM-CSF at Presentation
Description: as for outcome 2
Time Frame: 0 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 9.9 (10.6) | 4.5 (7.4)

6. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. GM-CSF at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 7.2 (8.2) | 2.8 (4.2)

7. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. GM-CSF at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 7.7 (9.5) | 3.1 (4.5)

8. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-6 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 2017.9 (5436.7) | 2513.3 (6423.3)

9. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-6 at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 492.0 (1557.3) | 305.6 (764.6)

10. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-6 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 119.0 (247.0) | 52.3 (72.7)

11. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CXCL10 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 453.1 (496.0) | 1073.3 (2240.0)

12. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CXCL10 at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 816.6 (1243.1) | 846.1 (1534.6)

13. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CXCL10 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 450.7 (626.2) | 324.4 (369.3)

14. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. Il-5 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 5.8 (5.6) | 15.6 (44.8)

15. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. Il-5 at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 4.9 (4.4) | 18.4 (55.5)

16. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. Il-5 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 5.0 (4.6) | 2.4 (3.9)

17. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IFN-a2 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 16.6 (27.7) | 5.6 (5.0)

18. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IFN-a2 at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 12.3 (18.5) | 4.2 (2.6)

19. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IFN-a2 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 11.0 (9.9) | 4.0 (3.5)

20. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-4 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 19.5 (22.1) | 9.0 (12.0)

21. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-4 at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 14.6 (15.2) | 5.5 (5.0)

22. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-4 at 24 Hours
Description: as for outcome 2
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 14.4 (21.3) | 7.1 (10.9)

23. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL3 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 127.2 (176.9) | 55.5 (55.4)

24. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL3 at 12 Hours
Description: Exploratory analysis to map mechanistic inflammatory response. Comparison of mean cytokine concentrations between allocation arms. Comparing at 12 hours from presentation.
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 95.7 (128.7) | 48.5 (63.5)

25. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL3 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 98.0 (96.0) | 35.1 (35.1)

26. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-10 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 748.1 (2170.0) | 715.3 (2130.6)

27. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-10 at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 620.8 (2275.7) | 47.2 (100.2)

28. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-10 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 362.8 (1326.1) | 5.3 (4.6)

29. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-12p70 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 24.2 (59.6) | 6.4 (8.5)

30. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-12p70 at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 34.8 (108.5) | 3.9 (4.4)

31. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IL-12p70 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 11.4 (19.5) | 3.0 (3.1)

32. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL20 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 1792.5 (2390.7) | 708.2 (526.3)

33. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL20 at 12 Hours
Description: as for outcome 2
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 555.4 (504.1) | 659.3 (942.2)

34. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL20 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 314.1 (228.3) | 276.7 (215.1)

35. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IFN-gamma at Presentation
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 172.1 (194.7) | 31.2 (29.4)

36. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IFN-gamma at 0 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 114.3 (113.2) | 29.8 (23.2)

37. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. IFN-gamma at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 99.7 (102.7) | 27.0 (39.5)

38. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CXCL8 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 203.3 (320.3) | 149.5 (286.6)

39. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CXCL8 at 12 Hours
Description: as for outcome 3
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 114.4 (189.3) | 70.9 (94.4)

40. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CXCL8 at 24 Hours
Description: as for outcome 2
Time Frame: 24 hours from baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 88.3 (95.8) | 39.4 (39.7)

41. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL4 at 0 Hours
Description: as for outcome 2
Time Frame: 0 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 11.0 (7.3) | 19.6 (30.2)

42. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL4 at 12 Hours
Description: as for outcome 2
Time Frame: 12 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 6.8 (3.8) | 13.6 (22.4)

43. Primary Outcome: Longitudinal Change Over Time in Cell Types and Pro and Anti Inflammatory Cytokines in Sepsis. CCL4 at 24 Hours
Description: as for outcome 4
Time Frame: 24 hours from presentation
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albumin | Crystalloid
Number analyzed (Participants) | 14 | 12
pg/mL | 6.1 (3.7) | 9.8 (11.8)

ADVERSE EVENTS:
Time Frame: Adverse events recorded for this study up to 24 hours from presentation
Description: This study collected adverse event data related to this study alone (and its procedures, i.e. venepuncture).
  The report of mortality is a reflection of the patient's clinical course and was deemed of no relation to study interventions (i.e. venepuncture).
  The main, linked, cited study (ABC Sepsis) collected and describes adverse events relevant to the main study and its interventions.
Arm/Group | Albumin | Balanced Crystalloid
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT04963569/Prot_000.pdf